CLINICAL TRIAL: NCT01351220
Title: Community Dissemination of an Evidence-based CRC Screening Intervention
Brief Title: Community Dissemination of an Evidence-based Colorectal Cancer (CRC) Screening Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: RSGT CPPB-119384
Record Dates: First submitted 2011-05-06; First posted 2011-05-10 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-02

CONDITIONS: Colon Cancer; Rectal Cancer
Keywords: CRC screening; Prevention and early detection of CRC; Filipino; Dissemination
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Basic dissemination (Active Comparator)
  Interventions: Behavioral: Educational program and FOBT kits
- Organizational dissemination (Active Comparator)
  Interventions: Behavioral: Educational program and FOBT kits, and technical assistance

INTERVENTIONS:
Behavioral: Educational program and FOBT kits — Subjects will participate in a CRC small group educational program and receive FOBT kits from community health advisors who have received a one-time training session.
  Arms: Basic dissemination
Behavioral: Educational program and FOBT kits, and technical assistance — In addition to subjects' receipt of a CRC small group educational program and FOBT kits, leadership training and technical support will be provided to the community health advisors and selected leaders and members of the organization.
  Arms: Organizational dissemination

SUMMARY:
Filipino Americans have lower rates of colorectal cancer (CRC) screening, later stage of diagnosis and poorer survival relative to other racial/ethnic groups. To address this disparity, the investigators developed a multi-component intervention to increase CRC screening and have determined its efficacy in a randomized trial (Maxwell,et. al., 2010). This study aims to determine how an intervention to increase CRC screening can best be integrated within the cultural norms and existing structures of churches and community based organizations (CBOs) with predominantly Filipino American membership to ensure broad dissemination to those in need of screening.

The investigators will provide our partner CBOs with resources and technical assistance, including training of community volunteers as health advisors, to enable them to promote CRC screening to their constituents. Using a scientifically rigorous research design, the investigators will compare two dissemination strategies: Basic dissemination which consists of a single kick-off event during which community health advisors will receive print materials and FOBT kits for distribution and training on how to conduct educational small-group sessions; and Organizational dissemination aimed at integrating CRC screening dissemination into organizational practices and processes that can be sustained after the end of the study. The study will be implemented in 20 CBOs and will train 100 community health advisors (CHAs). The impact of the two dissemination strategies will be comprehensively assessed by collecting data at the CBO level, from the CHAs and from 1000 Filipino American participants. The investigators will compare the proportion of Filipino American participants who obtain CRC screening by dissemination strategy, but the investigators will also assess how many are reached, if the intervention is implemented as planned, how CBOs support the screening efforts at their regular activities, and if CBOs and CHAs maintain their efforts over the 4 years of the study.

The investigators hypothesize that CBOs can implement evidence-based strategies to promote CRC screening and CHAs in the organizational dissemination arm will reach more participants and more screened participants than CHAs in the basic dissemination arm; and organizations in the organizational dissemination arm will adopt more CRC screening activities and maintain these better than organizations in the basic dissemination arm.

ELIGIBILITY:
Inclusion Criteria:

* Filipino American
* 50 to 75 years of age
* Must not have been diagnosed with CRC
* Must not be adherent to USPSTF CRC screening guidelines

Exclusion Criteria:

* Not Filipino American
* Younger than 50 or older than 75 years of age
* Have been diagnosed with CRC
* Adherent to USPSTF CRC screening guidelines

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1100 (Actual)
Dates: Start 2010-07; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in receipt of CRC screening at 6 months and 24 months | baseline, 6-month and 24-month post intervention
  Subjects will receive any one of the 3 recommended CRC screening tests namely, Fecal Occult Blood Test, Flexible sigmoidoscopy or Colonoscopy

SECONDARY OUTCOMES:
Change from Baseline in intention to obtain screening at 6 months and 24 months | baseline, 6-months and 24-months after exposure to the intervention
Change from Baseline in CRC screening knowledge at 6 months and 24 months | baseline, 6 months and 24 months after exposure to the educational program
Change from Baseline in frequency of patient provider communication at 6 months and 24 months | baseline, 6 and 24 months after exposure to the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Annette E Maxwell, Dr.P.H., Principal Investigator — University of California, Los Angeles; Leda L Danao, Ph.D., Study Director — University of California, Los Angeles
Locations (1):
- UCLA Division of Cancer and Prevention Research, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maxwell AE, Bastani R, Danao LL, Antonio C, Garcia GM, Crespi CM. Results of a community-based randomized trial to increase colorectal cancer screening among Filipino Americans. Am J Public Health. 2010 Nov;100(11):2228-34. doi: 10.2105/AJPH.2009.176230. Epub 2010 Sep 23. PMID 20864724
- [Derived] Maxwell AE, Crespi CM, Arce AA, Bastani R. Exploring the effects of longstanding academic-community partnerships on study outcomes: A case study. Prev Med Rep. 2017 Sep 12;8:101-107. doi: 10.1016/j.pmedr.2017.09.003. eCollection 2017 Dec. PMID 28948137
- [Derived] Maxwell AE, Danao LL, Cayetano RT, Crespi CM, Bastani R. Implementation of an evidence-based intervention to promote colorectal cancer screening in community organizations: a cluster randomized trial. Transl Behav Med. 2016 Jun;6(2):295-305. doi: 10.1007/s13142-015-0349-5. PMID 27282431